CLINICAL TRIAL: NCT04501432
Title: Cardiac Rehabilitation and Ongoing Physical Activity During the Coronavirus Disease (COVID-19) Pandemic: An Exploratory Mixed-Methods Study
Brief Title: Cardiac Rehabilitation and Ongoing Physical Activity During COVID-19
Acronym: CODIS
Status: Completed | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Collaborators: Institute of Sports Medicine, Prevention and Rehabilitation, Salzburg, Austria (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23_CODIS
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Rehabilitation
Keywords: COVID-19; Exercise Tolerance; Physical Activity; Qualitative Interview; Secondary Prevention; Social Distancing
MeSH Terms: conditions — COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Rehabilitation: Participants will be recruited from a group of patients who regularly attended group-based cardiac rehabilitation exercise training at the study site until COVID-19 restrictions (national lockdown) came into force on 16th March 2020.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study does not include an intervention

SUMMARY:
The current Coronavirus Disease 2019 (COVID-19) pandemic has resulted in extraordinary public health orders of social distancing and self-isolation, leading to widespread disruption and discontinuation of cardiac rehabilitation programmes and other social opportunities for cardiovascular disease (CVD) patients to exercise. In Austria, the government initiated drastic public health measures (national lockdown) on March 16, 2020, leading to closure of all outpatient cardiac rehabilitation facilities and restriction of inpatient rehabilitation to patients with urgent medical indications only.

This study aims to explore the impact of COVID-19-related national lockdown and public health restrictions on cardiac rehabilitation patients, with respect to maintenance of physical activity for secondary CVD prevention.

The study poses three research questions, which will be addressed in a mixed-methods study with sequential quantitative-qualitative (QUANT-QUAL) design:

1. What was the impact of the COVID-19-related lockdown on patients' physical activity and physical fitness levels? (QUANT stage)
2. What was the patient experience of the closure of group-based cardiac rehabilitation training due to COVID-19 public health restrictions? (QUAL stage)
3. Which insights and learning points may be drawn from patients' experiences during COVID-19 public health restrictions with respect to the provision of home-based digital support for physical activity? (QUAL stage)

The study will recruit a cohort of up to 40 cardiac rehabilitation patients from one outpatient cardiac rehabilitation centre in Salzburg, Austria, whose rehabilitation programme was interrupted by COVID-19 public health orders, including "lockdown".

Patients will undergo re-assessment of physical fitness in cycle ergometry test and re-assessment of cardiovascular risk profile. This will be compared with patients' most recent available test results from before the COVID-19 lockdown (i.e. prior to mid-March 2020) from patient records. Additionally, patients will take part in a semi-structured qualitative interview in which they will be invited to reflect on their personal experiences during the COVID-19 lockdown and thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and over)
* Cardiovascular disease (CVD)
* Currently enrolled in outpatient cardiac rehabilitation training at the study site
* Informed consent

Exclusion Criteria:

* Contraindications for cardiopulmonary exercise testing
* Pathologies limiting exercise performance
* Pregnancy or breastfeeding
* Limited German language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A group of patients who regularly attended group-based cardiac rehabilitation exercise training at the study site until COVID-19 restrictions (national lockdown) came into force on 16th March 2020.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Work load (W) | up to 12 months
  Maximal work load (W) achieved in cycle ergometry test
Work load % of predicted value | up to 12 months
  Maximal work load (W) achieved in cycle ergometry test expressed as percentage of predicted value
Heart rate (bpm) | up to 12 months
  Maximal heart rate (bpm) during cycle ergometry test
Framingham Recurrent Coronary Heart Disease risk score | up to 12 months
  Range 1% to 29%, higher percentage indicating worse risk estimate

SECONDARY OUTCOMES:
Metabolic Equivalent (MET) minutes / week | up to 12 months
  MET-minutes/week calculated from patient self-report of physical activity (International Physical Activity Questionnaire, IPAQ, 7 day version)
Patient Experience | 5 months
  Semi-structured qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Stefan T Kulnik, PhD MRes, Principal Investigator — Ludwig Boltzmann Institute for Digital Health and Prevention
Locations (1):
- Institute of Sports Medicine, Prevention and Rehabilitation, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No